CLINICAL TRIAL: NCT00000135
Title: Monoclonal Antibody CMV Retinitis Trial (MACRT)
Brief Title: Studies of the Ocular Complications of AIDS (SOCA)--Monoclonal Antibody CMV Retinitis Trial (MACRT)
Acronym: MACRT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-34
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections; Cytomegalovirus Retinitis
MeSH Terms: conditions — HIV Infections; Cytomegalovirus Retinitis | interventions — sevirumab; Antibodies, Monoclonal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSL-109 (Experimental): The dose MSL-109 administered by intravenous infusion every 2 weeks 60 mg.
  Interventions: Drug: MSL-109
- Placebo (Placebo Comparator): Placebo administered intravenous infusion every 2 weeks 60 mg.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MSL-109 — 60 mg, IV (in vein) every two weeks, treatment continued until death or common closeout.
  Other Names: Monoclonal antibodies
  Arms: MSL-109
Other: Placebo — 60 mg, IV (in vein) every two weeks, treatment continued until death or common closeout.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of a human anti-CMV monoclonal antibody, MSL-109, as adjunct therapy for controlling CMV retinitis.

DETAILED DESCRIPTION:
CMV retinitis is the most common intraocular infection in patients with AIDS and is estimated to affect 35 to 40 percent of patients with AIDS. Untreated CMV retinitis is a progressive disorder, the end result of which is total retinal destruction and blindness. As of September 1996, drugs approved by the United States Food and Drug Administration (FDA) for the treatment of CMV retinitis were ganciclovir (Cytovene), foscarnet (Foscavir), and cidofovir (Vistide). All systemically administered anti-CMV drugs are given in a similar fashion consisting of initial 2-week high-dose treatment (induction) to control the infection followed by long-term lower dose treatment (maintenance) to prevent relapse. Ganciclovir is available in both intravenous and oral formulations, foscarnet only in an intravenous formulation, and cidofovir is given by intermittent intravenous administration. A surgically implanted intraocular sustained-release ganciclovir device (Vitrasert) is also approved by the FDA for the treatment of CMV retinitis.

Despite the use of continuous maintenance therapy, given enough time, all patients with CMV retinitis on systemically administered drugs relapse. Preliminary studies suggested that the anti-CMV monoclonal antibody, MSL-109, when administered in conjunction with ganciclovir, markedly prolonged the time to relapse. Therefore, a randomized controlled clinical trial evaluating MSL-109 as adjunct therapy was conducted.

The MACRT was a randomized, placebo-controlled, multicenter clinical trial evaluating the efficacy and safety of MSL-109 as adjunct therapy for the treatment of CMV retinitis. Patients with CMV retinitis, both those newly diagnosed and those suffering a relapse with active retinitis, were eligible. Primary therapy (e.g., ganciclovir, foscarnet, etc.) was determined by the treating local physician. The patients enrolled in the trial were randomized to either MSL-109 or placebo, administered as a rapid intravenous infusion every 2 weeks. Outcomes included survival, retinitis progression, change in amount of retinal area involved by CMV, loss of visual function (acuity and field), and morbidity.

ELIGIBILITY:
Inclusion criteria:

* 13 years or older at entry
* Diagnosis of AIDS according to the Centers for Disease Control and Prevention (CDC) definition
* Diagnosis of active CMV retinitis as determined by a SOCA-certified ophthalmologist at time of enrollment
* At least one lesion whose size is one-quarter or more optic disc area
* Currently receiving (for relapsed patients) or scheduled to receive (for newly diagnosed patients) drugs for primary treatment of CMV retinitis that are not contraindicated for use with MSL-109
* Visual acuity, in at least one eye that meets other eligibility criteria, of 3 or more letters on ETDRS chart at 1 meter distance (Snellen equivalent 5/200). Patients with poorer visual acuity may be enrolled if the visual acuity impairment is possibly reversible (eg, due to optic disc edema) and vision is at least light perception in that eye
* Karnofsky score of 60 or more
* Willingness and ability, with the assistance of a caregiver if necessary, to comply with treatment and follow up procedures
* signed consent statement

Exclusion criteria:

* Current treatment with intravenous immune globulin (IVIG), CMV immune globulin (CMVIG), alpha-interferon (alpha-IFN), gamma-interferon (gamma-IFN) or interleukin-2 (IL-2)
* Media opacity that precludes visualization of the fundus in all eyes meeting eligibility criteria
* Active medical problems, including drug or alcohol abuse, that are considered sufficient to hinder compliance with treatment or follow up procedures
* Retinal detachment, not scheduled for surgical repair, in all eyes meeting other eligibility criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 1995-09; Primary Completion 1996-08 (Actual); Study Completion 1996-08 (Actual)

REFERENCES:
- [Result] MSL-109 adjuvant therapy for cytomegalovirus retinitis in patients with acquired immunodeficiency syndrome: the Monoclonal Antibody Cytomegalovirus Retinitis Trial. The Studies of Ocular Complications of AIDS Research Group. AIDS Clinical Trials Group. Arch Ophthalmol. 1997 Dec;115(12):1528-36. PMID 9400786
- [Result] Jabs DA, Gilpin AM, Min YI, Erice A, Kempen JH, Quinn TC; Studies of Ocular Complications of AIDS Research Group. HIV and cytomegalovirus viral load and clinical outcomes in AIDS and cytomegalovirus retinitis patients: Monoclonal Antibody Cytomegalovirus Retinitis Trial. AIDS. 2002 Apr 12;16(6):877-87. doi: 10.1097/00002030-200204120-00007. PMID 11919489
- [Result] Davidson M, Min YI, Holbrook JT, Van Natta M, Quinn TC, Murphy RL, Welch W, Jabs DA, Meinert CL; Studies of Ocular Complications of AIDS Research Group. Influence of filgrastim (granulocyte colony-stimulating factor) on human immunodeficiency virus type 1 RNA in patients with cytomegalovirus retinitis. J Infect Dis. 2002 Oct 1;186(7):1013-8. doi: 10.1086/342956. Epub 2002 Aug 29. PMID 12232843
- [Result] Gilpin AM, Holbrook JT, Jabs DA, Meinert CL; Studies of Ocular Complications of AIDS Research Group. Data and safety monitoring board deliberations resulting in the early termination of the Monoclonal Antibody Cytomegalovirus Retinitis Trial. Control Clin Trials. 2003 Feb;24(1):92-8. doi: 10.1016/s0197-2456(02)00268-4. PMID 12559647
- [Derived] Holland GN, Van Natta ML, Goldenberg DT, Ritts R Jr, Danis RP, Jabs DA; Studies of Ocular Complications of AIDS Research Group. Relationship Between Opacity of Cytomegalovirus Retinitis Lesion Borders and Severity of Immunodeficiency Among People With AIDS. Invest Ophthalmol Vis Sci. 2019 May 1;60(6):1853-1862. doi: 10.1167/iovs.18-26517. PMID 31042791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization was stratified on the basis of whether patients had untreated or relapsed retinitis. Primary drug therapy for CMV retinitis was determined by the treating physician.
Pre-assignment Details: Two hundred and nine patients with acquired immunodeficiency syndrome and active CMV retinitis were enrolled in a multicenter, phase 2/3, randomized, placebo controlled clinical trial. Patients received adjuvant treatment with MSL-109, 60mg intravenously every 2 weeks, or placebo,.
Groups:
- Placebo: Placebo administered intravenous infusion every 2 weeks 60 mg.
  MSL-109: 60 mg, IV (in vein) every two weeks, treatment continued until death or common closeout.
Period: Overall Study
Arm/Group | MSL-109 | Placebo
Started | 104 | 105
Completed | 77 | 91
Not Completed | 27 | 14
Not completed — Death | 27 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSL-109 | Placebo | Total
Number analyzed (Participants) | 104 | 105 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 104 | 105 | 209
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 93 | 94 | 187
Region of Enrollment [Number; unit: participants]
  United States | 104 | 105 | 209

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rate
Description: to evaluate the efficacy of an intravenous human monoclonal antibody to cytomegalovirus (CMV), MSL-109, as adjuvant treatment for CMV retinitis. .
Time Frame: All patients enrolled were followed for a 17 month period or until a common study closing date
Measure: Number; unit: deaths per person-year
Arm/Group | MSL-109 | Placebo
Number analyzed (Participants) | 104 | 105
deaths per person-year | 0.68 | 0.31

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | MSL-109 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/105
Other Adverse Events (participants affected / at risk) | 0/104 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other